CLINICAL TRIAL: NCT06241430
Title: Hemodynamic-Guided Optimization With the CardioMEMS Device of Patients With Heart Failure and Secondary Mitral Regurgitation Undergoing Mitral Transcatheter Edge-to-Edge Repair With the MitraClip Device
Brief Title: The CardioClip Study
Acronym: CardioClip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Nir Uriel, Seymour, Paul, and Gloria Milstein Professor of Cardiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU9731
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Mitral Regurgitation
Keywords: Heart failure; Reduced ejection fraction; Mitral regurgitation; mTEER (mitral transcatheter edge-to-edge repair); CardioMems (implantable pulmonary artery pressure sensor); Guideline-directed medical therapy (GDMT); HF hospitalization (HFH); Clinical trial; Hemodynamic monitoring; Cardiovascular outcomes
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: Evaluating the effect of hemodynamic-guided GDMT titration with CardioMems on HFH in individuals with functional MR and HF undergoing mTEER, compared to usual care involving GDMT.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CardioMems (Experimental): Participants randomized to this arm will receive hemodynamic-guided GDMT titration with CardioMems.
  Interventions: Device: CardioMEMS
- Usual Care (No Intervention): Participants randomized to this arm will receive usual care involving GDMT.

INTERVENTIONS:
Device: CardioMEMS — Hemodynamic-guided optimization will be performed using the CardioMEMS CardioClip device.
  Arms: CardioMems

SUMMARY:
The CardioClip study is exploring the use of a wireless sensor to monitor pressure in the pulmonary artery. This sensor is inserted much like the mTEER procedure, a non-surgical method through a vein in the groin. The investigators want to find out if the sensor, by constantly sending information about heart function, can help improve patient outcomes. This means doctors could adjust medications based on real-time pressure changes detected by the sensor. The results from this study will help pave the way for future trials, asking if using these wireless sensors could benefit people with valve disease and heart failure.

DETAILED DESCRIPTION:
Patients with heart failure suffer considerably. They experience an increased risk of death and are hospitalized with symptoms of heart failure frequently. Often times, heart failure results in abnormal function of the mitral valve (one of the key valves separating the heart's main pumping chamber - the left ventricle - from the left atrium, which collects oxygenated blood from arteries in the lung). This abnormal function causes the valve to leak - a condition called mitral regurgitation - that perpetuates and can exacerbate heart failure.

Recently, researchers have developed a procedure for patients with mitral regurgitation in the setting of heart failure called mitral transcatheter edge-to-edge repair (mTEER). In this procedure, a "clip" is deployed to grasp the mitral valve leaflet and re-approximate them, thereby reducing the amount of mitral regurgitation. This procedure is performed by accessing one of the large veins in the body and no surgical intervention is required. Patients typically recover within 24 hours and are discharged home without the prolonged recovery periods associated with traditional therapies for mitral regurgitation like open heart surgery and mitral valve repair or replacement. Moreover, the procedure is exceedingly safe, with a very low risk of significant adverse complications.

While mTEER reduces the risk of death and hospitalization for heart failure compared with the standard of care (i.e., medicines geared at improving heart function), many patients still suffer significant adverse events within a five year period. Accordingly, the investigators are interested in identifying strategies to further improve outcomes for patients with heart failure and significant mitral regurgitation. The CardioClip study endeavors to use another technology - a wireless pulmonary artery pressure sensor - that is implanted in a similar fashion to the way mTEER is performed (i.e., percutaneously, without surgery, through one of the veins in the groin), to see whether clinical outcomes can be improved further. The sensor continuously transmits information regarding heart function to clinicians who can optimize medications and their doses according to dynamic changes in pressure noted by the sensor.

ELIGIBILITY:
Inclusion Criteria:

* Significant (moderate-severe [3+] or severe [4+] secondary MR)
* Left ventricular dysfunction (ejection fraction >20% and <50%)
* New York Heart Association (NYHA) class II-IVa symptoms
* Sign informed consent to participate in the study

Exclusion Criteria:

* Left ventricular (LV) end-systolic dimension 70 mm
* PA systolic pressure 70 mmHg (fixed)
* Mitral valve (MV) orifice area <4.0 cm2
* Commissural MR jet or leaflet anatomy not suitable for mTEER
* Likely to undergo heart transplantation or LV assist device implantation in the next 12 months
* Recurrent (i.e., >1) pulmonary embolism or deep vein thrombosis
* Complex congenital heart disease
* Mechanical right heart valve (tricuspid or pulmonic)
* Cardiac resynchronization therapy implanted within 3 months of enrollment
* Hypersensitivity to aspirin and/or clopidogrel
* History of medication non-adherence

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary (OS) score between baseline (pre-mTEER) and 12 months after mTEER. | 12 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. To facilitate interpretation, all scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life (i.e., higher score indicates a better outcome). The Overall Summary (OS) score is the mean of four subdomain scores, each ranging from 0 to 100. A higher OS score indicates better outcome.

SECONDARY OUTCOMES:
All-cause mortality rate at 12 months | 12 months
  All-cause mortality rate will be calculated at 12 months.
Rate of HFH at 12 months | 12 months
  Heart failure hospitalization (HFH) rate will be calculated.
Number of participants who achieve excellent clinical outcome | 12 months
  An excellent clinical outcome is defined by a) survival, b) KCCQ-OS >60 points, and c) no decline ≥10 points in the KCCQ-OS relative to baseline at 12 months
KCCQ score - Physical Function domain | Baseline, 1 month, 6 months, 12 months post-mTEER
  The KCCQ-OS evaluates health status from four principal domains: physical function, social function, symptoms, and quality of life. Participants receive a score for 0 to 100 in each domain, with higher scores indicating better health status in that specific domain. The score for each domain will be an individual secondary endpoint.
KCCQ score - Social Function domain | Baseline, 1 month, 6 months, 12 months post-mTEER
  The KCCQ-OS evaluates health status from four principal domains: physical function, social function, symptoms, and quality of life. Participants receive a score for 0 to 100 in each domain, with higher scores indicating better health status in that specific domain. The score for each domain will be an individual secondary endpoint.
KCCQ score - Symptoms domain | Baseline, 1 month, 6 months, 12 months post-mTEER
  The KCCQ-OS evaluates health status from four principal domains: physical function, social function, symptoms, and quality of life. Participants receive a score for 0 to 100 in each domain, with higher scores indicating better health status in that specific domain. The score for each domain will be an individual secondary endpoint.
KCCQ score - Quality of Life domain | Baseline, 1 month, 6 months, 12 months post-mTEER
  The KCCQ-OS evaluates health status from four principal domains: physical function, social function, symptoms, and quality of life. Participants receive a score for 0 to 100 in each domain, with higher scores indicating better health status in that specific domain. The score for each domain will be an individual secondary endpoint.
Change in New York Heart Association (NYHA) Classification at 1-, 6-, and 12-months post-mTEER relative to baseline. | Baseline, 1 month, 6 months, 12 months
  The different classes in the NYHA Classification of Heart Failure are:
  Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
6-minute walk test (6MWT) at 12 months | 12 months
  The 6 minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance. The score of the test is the distance a patient walks in 6 minutes at 12 months.
Change in 6-minute walk test (6MWT) from baseline to 12 months | Baseline and 12 months
  The 6 minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance. The score of the test is the distance a patient walks in 6 minutes. Change of score at baseline and then at 12 months will be calculated.
Win ratio | Baseline and 12 months
  Win ratio for the hierarchical endpoint of KCCQ improvement ≥10 points at 12 months, NYHA functional class improvement ≥1 class at 12 months, 6MWT improvement ≥30 meters at 12 months, HFH at 12 months, and all-cause mortality at 12 months.
Echocardiographic estimates of RV-PA coupling indices | 12 months
  Right ventricular (RV)-pulmonary arterial (PA) (RV-PA) coupling indices will be measured (mm/mmHg) will be measured to determine how the right ventricle and pulmonary circulation interact.
Device-related (MitraClip) complications at 12 (single-leaflet device detachment, device embolization, endocarditis requiring surgery, mitral stenosis requiring surgery) | 12 months
  MitraClip complications
Single-leaflet Device Detachments | 12 months
  Device-related MitraClip complications: Total number of single-leaflet device detachment events.
Device Embolizations (MitraClip) | 12 months
  Device-related MitraClip complications: Total number of device embolizations.
Endocarditis (Requiring Surgery) | 12 months
  Device-related MitraClip complications: Total number of endocarditis events requiring surgery.
Mitral Stenosis (Requiring Surgery) | 12 months
  Device-related MitraClip complications: Total number of mitral stenosis events requiring surgery.
Device- or System-related Failures | 12 months
  Device-related CardioMEMS complications: Total number of device- or system-related failures.
In Situ Pulmonary Thrombosis | 12 months
  Device-related CardioMEMS complications: Total number of in situ pulmonary thrombosis.
Device Embolizations (CardioMEMS) | 12 months
  Device-related CardioMEMS complications: Total number of device embolizations

CONTACTS AND LOCATIONS:
Overall Officials: Nir Uriel, MD, Principal Investigator — Columbia University; Michael Brener, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No